CLINICAL TRIAL: NCT04462497
Title: Chest-Up: Obtaining Safe Positioning for Thoracic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019/00637
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-06

CONDITIONS: Thoracic
Keywords: Intraoperative; Lateral decubitus

STUDY DESIGN:
Intervention Model Description: There will be 2 groups of a patients randomized to either the existing method of head support (sponge and towel stack) or prototype head and neck support device.
Who Masked: Participant
Masking Description: One group of patients will receive the existing method of head support (control group), the other group will receive the prototype head and neck support device (study group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants will receive the existing method of head support (sponge and towel stack) intraoperatively.
- Study Group (Experimental): Participants will receive the prototype head and neck support device intraoperatively.
  Interventions: Other: Prototype device

INTERVENTIONS:
Other: Prototype device — Patients will receive the prototype head and neck support device to be used intraoperatively.
  Arms: Study Group

SUMMARY:
Thoracotomy surgeries, both open and video assisted, are often carried out in the lateral decubitus position to optimize surgical access to the operative side. However, this position is also associated with mechanical injuries of the shoulder joint ligaments and pulling on the structures of the brachial plexus. The neck is laterally flexed and has potential to cause mechanical injury as well due to the dependent position of the patient's head.

The current method of positioning involves stacking of towels under a head support. To the study team's knowledge, no pre-formed head and neck support exists that can cope with the required surgical position. Thus, the study team has conceptualized an adaptive head and neck support pillow to meet this need and address patient safety concerns.

DETAILED DESCRIPTION:
Thoracotomy surgeries, both open and video assisted, are often carried out in the lateral decubitus position. This necessitates the flexion of the surgical table into an inversed 'v' shape to optimize surgical access to the operative side.

However, this position is also associated with mechanical injuries of the shoulder joint ligaments and pulling on the structures of the brachial plexus. With the dependent position of the patient's head, the neck is laterally flexed and has potential to cause mechanical injury as well. Normal cervical flexion range of motion is about 20-45 degrees, although this may be restricted in patients with cervical spine pathology or in the elderly. Ipsilateral shoulder pain (ISP) post thoracic surgery is a recognized complication and can be difficult to treat. While referred pain from the phrenic nerve is the well-studied cause, some literature noted that ipsilateral shoulder pain of the musculoskeletal type is more intense than referred ipsilateral shoulder pain. Rarer complications are not well reported but may include paraplegia and winging of the scapula. Positioning is also more challenging in obese patients, accompanied by a higher risk of position related complications.

The current method of positioning involves stacking of towels under a head support. To the study team's knowledge, no pre-formed head and neck support exists that can cope with the required surgical position, movements during the flexing and unflexing of the surgical table, as well as the different physical attributes of different patients.

The study team is concerned regarding the inherent dangers to patient safety, such as slippage or instability of a stack of towels, and the need for at least 3 personnel to help support the patient's head and neck adequately during positioning. With the anaesthetist preoccupied with holding the patient's head during positioning, there is the potential for inattention to other important issues such as haemodynamic changes. Existing methods of using a bean bag have fallen out of favor in our institution due to restriction of surgical access, bulkiness of the bean bag, need for a suction pump, and risk of pressure injury. The bean bag's main application is for maintaining the body in a lateral position, not for head and neck support.

Hence, the study team conceptualized the adaptive head and neck support pillow to meet this need and address patient safety concerns. Beyond thoracic surgery, it is hoped it will have applications in other situations requiring lateral decubitus positioning with flexion of the surgical table, such as nephrectomies.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years and above
* Listed for elective thoracic surgery in the lateral decubitus position

Exclusion Criteria:

* Patient refusal
* Age below 21 years
* Emergency cases
* Pregnant patients
* Cognitively impaired patients
* Unconscious patients

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-07-23 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Degrees of flexion during positioning | Intraoperatively
  During positioning of patient, the goniometer will be used to measure and record the degree of lateral neck movement during the positioning process. Degrees of deviation from the maximum comfortable degree of the patient's lateral flexion calculated.

SECONDARY OUTCOMES:
Post-operative follow-up | Postoperative days 1 and 2
  Patient will be contacted on postoperative day 1 and 2 to ask about neck or shoulder pain, numbness or weakness.
User Satisfaction | Immediate postoperative
  Gather user satisfaction feedback from surgeons and anaesthetists regarding usability and satisfaction using a Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Xian Li Deborah Khoo, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blichfeldt-Eckhardt MR, Andersen C, Ording H, Licht PB, Toft P. Shoulder Pain After Thoracic Surgery: Type and Time Course, a Prospective Cohort Study. J Cardiothorac Vasc Anesth. 2017 Feb;31(1):147-151. doi: 10.1053/j.jvca.2016.04.032. Epub 2016 May 9. PMID 27576216
- [Background] Yousefshahi F, Predescu O, Colizza M, Asenjo JF. Postthoracotomy Ipsilateral Shoulder Pain: A Literature Review on Characteristics and Treatment. Pain Res Manag. 2016;2016:3652726. doi: 10.1155/2016/3652726. Epub 2016 Nov 28. PMID 28018130
- [Background] Bhuiyan MS, Mallick A, Parsloe M. Post-thoracotomy paraplegia coincident with epidural anaesthesia. Anaesthesia. 1998 Jun;53(6):583-6. doi: 10.1046/j.1365-2044.1998.00470.x. PMID 9709146
- [Background] Martin JT. Postoperative isolated dysfunction of the long thoracic nerve: a rare entity of uncertain etiology. Anesth Analg. 1989 Nov;69(5):614-9. PMID 2552867